CLINICAL TRIAL: NCT03111108
Title: A Multi-Site, Open-Label, Partially-Randomized Trial of the Efficacy and Safety of Fixed Dose Elbasvir/Grazoprevir (EBR/GZR) Based Regimens in French Subjects With Chronic Hepatitis C Virus (HCV) Genotype 4 Infection
Brief Title: Efficacy and Safety of Elbasvir (MK-8742) + Grazoprevir (MK-5172) in Treatment-Naïve/Treatment-Experienced (TN/TE) French Participants With Hepatitis C Virus (HCV) Genotype 4 (GT4) Infection (MK-5172-096)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5172-096; 2016-001159-37 (EudraCT Number); MK-5172-096 (Other: Merck Protocol Number)
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Results first posted 2019-11-12 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Hepatitis C Virus (HCV) Infection
MeSH Terms: conditions — Hepatitis C; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: EBR/GZR for 8 Weeks (Experimental): Treatment-naïve participants with stage 0-2 fibrosis (F0-F2) receive FDC of EBR/GZR (50 mg/100 mg) for 8 weeks, with 24 weeks of follow-up.
  Interventions: Drug: EBR/GZR (50 mg/100 mg) FDC
- Arm 2: EBR/GZR for 12 Weeks (Experimental): Treatment-naïve participants with F0-F2 stage fibrosis, treatment-naïve participants with F3-F4 stage fibrosis, and treatment-experienced participants with F0-F4 stage fibrosis receive FDC of EBR/GZR (50 mg/100 mg) for 12 weeks, with 24 weeks of follow-up.
  Interventions: Drug: EBR/GZR (50 mg/100 mg) FDC

INTERVENTIONS:
Drug: EBR/GZR (50 mg/100 mg) FDC — One FDC tablet taken once daily by mouth for 8 or 12 weeks depending upon randomization.
  Other Names: MK-5172A

SUMMARY:
The purpose of this study was to evaluate the efficacy of 8 and 12 weeks of treatment with a fixed dose combination (FDC) of elbasvir (EBR) 50 mg + grazoprevir (GZR) 100 mg (i.e., MK-5172A) as assessed by the percentage of participants with hepatitis C virus (HCV) genotype (GT) 4 infection that achieve sustained virologic response (HCV ribonucleic acid [RNA] < Lower Limit of Quantification [LLOQ]) 12 weeks after the end of study therapy (SVR12). This study also evaluated the safety and tolerability of EBR/GZR.

ELIGIBILITY:
Inclusion Criteria:

* Be a current resident of France
* Have HCV RNA (≥ 10,000 IU/mL in peripheral blood) at the time of screening
* Have documented chronic HCV GT4 (with no evidence of non-typeable or mixed genotype) infection
* Have liver biopsy performed within 24 months of Day 1 of this study (if participant has cirrhosis, there is no time restriction on biopsy), or have FibroScan® performed within 12 months of Day 1 of this study with interpretable result in kilopascals (kPa) as follows: Fibrosis score of F0-F2, Fibrosis score of F3, or Cirrhosis (F4)
* Have a prior treatment history of either HCV TN or HCV TE with interferon (IFN) +/- ribavirin (RBV) +/- Sofosbuvir (SOF) (on-treatment failure, relapser, or other/intolerant)
* Females who are of reproductive potential must agree to avoid becoming pregnant while receiving study drug and for 14 days after the last dose of study drug by complying with one of the following: (1) practice abstinence from heterosexual activity OR (2) use (or have her partner use) acceptable contraception during heterosexual activity
* If Human Immunodeficiency Virus (HIV) co-infected, then have HIV-1 infection documented prior to screening

Exclusion Criteria:

* Had prior treatment (defined as 1 dose or more) with direct-acting antiviral (DAA) therapy
* Has evidence of decompensated liver disease manifested by the presence of or history of ascites, esophageal or gastric variceal bleeding, hepatic encephalopathy, or other signs or symptoms of active advanced liver disease
* Classified as Child-Pugh B or C or has a Child Pugh-Turcotte score (CPT) > 6
* Has cirrhosis and liver imaging within 6 months of Day 1 showing evidence of hepatocellular carcinoma (HCC) or is under evaluation for HCC
* Hepatitis B virus surface antigen (HBsAg) positive at screening. Participants who are HBsAg negative and hepatitis B core antibody (anti-HBc) positive at screening may be included
* Under evaluation for active or suspected malignancy, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer Currently participating or has participated in a study with an investigational compound within 30 days of signing informed consent and is not willing to refrain from participating in another such study during the course of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (13):
- France (13):
  - CHU Amiens-Picardie - Hopital Sud ( Site 0217), Amiens
  - CHU Jean Minjoz ( Site 0213), Besançon
  - CHU Henri Mondor ( Site 0206), Créteil
  - CHU de Grenoble - Hopital Michallon ( Site 0208), Genoble
  - CHU Dupuytren ( Site 0209), Limoges
  - Hopital Saint Eloi ( Site 0207), Montpellier
  - C.H.U. de Nice Hopital de l Archet 2 ( Site 0215), Nice
  - Centre Hospitalier Regional du Orleans ( Site 0212), Orléans
  - Hopital Beaujon ( Site 0201), Paris
  - Hopital Cochin ( Site 0211), Paris
  - Hopital Saint Antoine ( Site 0200), Paris
  - CHU de Toulouse - Hopital Purpan ( Site 0216), Toulouse
  - CHU de Nancy Hopital Brabois Adultes ( Site 0204), Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Asselah T, Pol S, Hezode C, Loustaud-Ratti V, Leroy V, Ahmed SNS, Ozenne V, Bronowicki JP, Larrey D, Tran A, Alric L, Nguyen-Khac E, Robertson MN, Hanna GJ, Brown D, Asante-Appiah E, Su FH, Hwang P, Hall JD, Guidoum A, Hagen K, Haber BA, Talwani R, Serfaty L. Efficacy and safety of elbasvir/grazoprevir for 8 or 12 weeks for hepatitis C virus genotype 4 infection: A randomized study. Liver Int. 2020 May;40(5):1042-1051. doi: 10.1111/liv.14313. Epub 2020 Mar 22. PMID 31765046

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult male and female participants with chronic hepatitis C virus (HCV) genotype 4 (GT4) infection were enrolled at 12 study centers in France.
Groups:
- Arm 1: EBR/GZR for 8 Weeks: Treatment-naïve HCV GT4 participants with stage 0-2 fibrosis (F0-F2) received elbasvir/grazoprevir (EBR/GZR) fixed dose combination (FDC) [50 mg/100 mg] for 8 weeks, followed by 24 weeks of follow-up.
- Arm 2: EBR/GZR for 12 Weeks: Treatment-naïve HCV GT4 participants with F0-F2 stage fibrosis, treatment-naïve participants with F3-F4 stage fibrosis, and treatment-experienced participants with F0-F4 stage fibrosis received EBR/GZR FDC (50 mg/100 mg) for 12 weeks, followed by 24 weeks of follow-up.
Period: Overall Study
Arm/Group | Arm 1: EBR/GZR for 8 Weeks | Arm 2: EBR/GZR for 12 Weeks
Started | 53 | 64
Completed | 52 | 63
Not Completed | 1 | 1
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: EBR/GZR for 8 Weeks: Treatment-naïve HCV GT4 participants with stage 0-2 fibrosis (F0-F2) received EBR/GZR FDC (50 mg/100 mg) for 8 weeks, followed by 24 weeks of follow-up.
- Total: Total of all reporting groups
Arm/Group | Arm 1: EBR/GZR for 8 Weeks | Arm 2: EBR/GZR for 12 Weeks | Total
Number analyzed (Participants) | 53 | 64 | 117
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.5 (12.9) | 56.0 (9.7) | 54.0 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 32 | 61
  Male | 24 | 32 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 29 | 49
  White | 28 | 29 | 57
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response 12 Weeks After End of Treatment (SVR12)
Description: The percentage of participants to achieve SVR12 was determined for each arm (SVR12 was defined as HCV ribonucleic acid [RNA] < lower limit of quantification [LLOQ] at 12 weeks after the end of all study therapy). Plasma HCV RNA was measured using the COBAS™ AmpliPrep/COBAS™ TaqMan HCV Test, v2.0®, which has a LLOQ of 15 IU/mL.
Time Frame: 12 weeks after completing study treatment (Arm 1: Week 20 / Arm 2: Week 24)
Population: All randomized participants who received ≥1 dose of study treatment are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Arm 1: EBR/GZR for 8 Weeks: Treatment-naïve HCV GT4 participants with stage 0-2 fibrosis (F0-F2) received EBR/GZR fixed dose combination (FDC) [50 mg/100 mg] for 8 weeks, followed by 24 weeks of follow-up.
Arm/Group | Arm 1: EBR/GZR for 8 Weeks | Arm 2: EBR/GZR for 12 Weeks
Number analyzed (Participants) | 53 | 64
Percentage of Participants | 94.3 [84.3 to 98.8] | 95.3 [86.9 to 99.0]

2. Primary Outcome: Number of Participants With ≥ 1 Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 14 weeks
Population: All randomized participants who received ≥1 dose of study treatment are included, classified according to treatment duration actually received.
Measure: Number; unit: Participants
Arm/Group | Arm 1: EBR/GZR for 8 Weeks | Arm 2: EBR/GZR for 12 Weeks
Number analyzed (Participants) | 53 | 64
Participants | 33 | 46

3. Primary Outcome: Number of Participants Who Discontinued From Study Treatment Due to an AE
Description: as for outcome 2
Time Frame: Up to Study Week 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Arm 1: EBR/GZR for 8 Weeks | Arm 2: EBR/GZR for 12 Weeks
Number analyzed (Participants) | 53 | 64
Participants | 0 | 0

4. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response 24 Weeks After End of Treatment (SVR24)
Description: The percentage of participants to achieve SVR24 was determined for each arm (SVR24 was defined as HCV RNA < LLOQ at 24 weeks after the end of all study therapy). Plasma HCV RNA was measured using the COBAS™ AmpliPrep/COBAS™ TaqMan HCV Test, v2.0®, which has a LLOQ of 15 IU/mL.
Time Frame: 24 weeks after completing study treatment (Arm 1: Week 32 / Arm 2: Week 36)
Population: All randomized participants who received ≥1 dose of study treatment are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm 1: EBR/GZR for 8 Weeks | Arm 2: EBR/GZR for 12 Weeks
Number analyzed (Participants) | 53 | 64
Percentage of Participants | 94.3 [84.3 to 98.8] | 93.8 [84.8 to 98.3]

5. Secondary Outcome: Prevalence of Baseline NS3 Resistance-Associated Substitutions (RASs) to EBR or GZR
Description: Blood samples for viral resistance assays were collected at Baseline (Day 1) and analyzed for substitutions in the NS3 gene region. Results are pooled for all participants with baseline sequencing data available, and the number of participants with RASs is reported according HCV genotype. Resistance-associated substitutions are defined as amino acid substitutions that confer reduced susceptibility to a direct-acting antiviral (DAA) and may contribute to virologic failure. The prevalence of baseline substitutions in participants infected with HCV GT4 subtypes was assessed by evaluating amino acid substitutions in NS3.
Time Frame: Day 1
Population: All randomized participants with baseline sequencing data for NS3 are included.
Measure: Number; unit: Participants
Arm/Group | Arm 1: EBR/GZR for 8 Weeks | Arm 2: EBR/GZR for 12 Weeks
Number analyzed (Participants) | 51 | 59
Participants
  GT4 | 5 | 6
  GT4D | 3 | 3
  GT4-Other | 6 | 9

6. Secondary Outcome: Prevalence of Baseline NS5A RASs to EBR or GZR
Description: Blood samples for viral resistance assays were collected at Baseline (Day 1) and analyzed for substitutions in the NS5A gene region. Results are pooled for all participants with baseline sequencing data available, and the number of participants with RASs is reported according HCV genotype. Resistance-associated substitutions are defined as amino acid substitutions that confer reduced susceptibility to a DAA and may contribute to virologic failure. The prevalence of baseline substitutions in participants infected with HCV GT4 subtypes was assessed by evaluating amino acid substitutions in NS5A.
Time Frame: Day 1
Population: All randomized participants with baseline sequencing data for NS5A are included.
Measure: Number; unit: Participants
Arm/Group | Arm 1: EBR/GZR for 8 Weeks | Arm 2: EBR/GZR for 12 Weeks
Number analyzed (Participants) | 53 | 63
Participants
  GT4 | 3 | 2
  GT4D | 10 | 16
  GT4-Other | 13 | 21

ADVERSE EVENTS:
Time Frame: Up to 36 weeks
Description: All participants who received ≥1 dose of study medication are included.
Arm/Group | Arm 1: EBR/GZR for 8 Weeks | Arm 2: EBR/GZR for 12 Weeks
All-Cause Mortality (participants affected / at risk) | 0/53 | 1/64
Serious Adverse Events (participants affected / at risk) | 2/53 | 2/64
Other Adverse Events (participants affected / at risk) | 27/53 | 38/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: EBR/GZR for 8 Weeks (N=53) | Arm 2: EBR/GZR for 12 Weeks (N=64)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: EBR/GZR for 8 Weeks (N=53) | Arm 2: EBR/GZR for 12 Weeks (N=64)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 3 (4)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (5)
Asthenia (General disorders) | 12 (12) | 14 (14)
Fatigue (General disorders) | 1 (1) | 4 (4)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 4 (4)
Nasopharyngitis (Infections and infestations) | 1 (1) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 3 (4) | 1 (1)
Headache (Nervous system disorders) | 9 (10) | 16 (16)
Insomnia (Psychiatric disorders) | 2 (2) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT03111108/Prot_SAP_000.pdf